CLINICAL TRIAL: NCT07284680
Title: Bio-implant Root Analogue Versus Conventional Screw-type Implant for Management of Pier Abutment in Mandibular Distal Extension Cases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hosam eldin Hegazy Mohamed Ebrahim Eid, postgrad student (master of prosthodontics), Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A11061222
Record Dates: First submitted 2025-11-23; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Implant Assesment
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioimolant (Experimental): bioimplant assessement
  Interventions: Device: Implant
- screw type conventional implant (Experimental): conventional screw type implant assessement
  Interventions: Device: Implant

INTERVENTIONS:
Device: Implant — construction of prothesis related to bioimplant or conventional implant

SUMMARY:
reviewing literature was lacking for bio implant and management of pier abutment in distal extension bases for this reason the aim of this research will be to use the bio implant in the management of pier abutment cases for distal extension denture base cases Aim of the study the aim of this study was to evaluate and compare the bioimplant root analogue implant with the conventional screw type implant the evaluation was done 0,3 and 6months of definitive prosthesis insertion regarding the following

1. radiographic evaluation of the alveolar bone hight as related to the bio implant ,conventional screw implant , pier abutment and RPD abutments : this will be done using standardized periapical digital radiographs
2. soft tissue evaluatins related to the bio implant ,conventional screw implant , pier abutment and RPD abutments this will be done using : A . modified plaque index (MPI) B . modified gingival index (MGI) C . peridontal pocket depth

ELIGIBILITY:
Inclusion Criteria:

* The patients had bilateral mandibular free-end partially edentulous cases with a pier abutment or a planned presence of pier abutment.
* The edentulous space mesial to the pier abutment has a hopeless tooth or root that was used for bio-implant insertion or conventional screw-type implants.
* Healthy patients with no systemic disease that can affect the implant surgery. This was verified by medical history in addition to a report from the physician.
* The patients have had dentulous maxillary jaw and mandibular free-end saddle for at least 6 months.
* Class I maxillo-mandibular relationship with adequate inter-arch distance.

Exclusion Criteria:

* Patients with metabolic disorders that affect osseointegration such as uncontrolled diabetes mellitus, immune disorders, and osteoporosis.
* Patients with heavy smoking habit
* Patients complaining of severe temporomandibular joint disorder.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
bone changes and soft tissue changes | after 3 and 6 months of denture insertion
  peri-implant bone and soft tissue changes and abutment teeth bone and soft tissue changes changes periapical X-ray for measurement of bone changes by millimeter periodontal probe for measurement of soft tissue changes by millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt